CLINICAL TRIAL: NCT00609830
Title: Osteoporosis Prevention Among People With Rheumatoid Arthritis Receiving Oral Glucocorticoid Therapy
Brief Title: GIOP Prevention Among People With Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Susan J. Blalock, PhD, The University of North Carolina at Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Arthritis Foundation
Record Dates: First submitted 2008-01-24; First posted 2008-02-07 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2008-01

CONDITIONS: Osteoporosis; Rheumatoid Arthritis
Keywords: Glucocorticoids; Osteoporosis; Rheumatoid Arthritis; Prevention; GIOP; Patient Education
MeSH Terms: conditions — Osteoporosis; Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (4):
- Tailored Materials (Experimental)
  Interventions: Behavioral: Tailored Materials
- Physician Feedback (Experimental)
  Interventions: Behavioral: Tailored Materials Plus Physician Feedback
- Generic Materials (Active Comparator)
  Interventions: Behavioral: Generic Materials
- Placebo Comparator (Placebo Comparator): Participants receive no information
  Interventions: Behavioral: No Information

INTERVENTIONS:
Behavioral: Tailored Materials — Participants received written educational materials concerning each behavior targeted. The materials were tailored to the participants' stage of change with respect to each behavior.
  Arms: Tailored Materials
Behavioral: Tailored Materials Plus Physician Feedback — Participants received written educational materials concerning each behavior targeted. The materials were tailored to the participant's stage of change with respect to each behavior. In additon, the participant's physician received information concerning the participant's status on each behavior targeted.
  Arms: Physician Feedback
Behavioral: Generic Materials — Participants received generic written educational materials about osteoporosis prevention.
  Arms: Generic Materials
Behavioral: No Information — Participants received no informational materials.
  Arms: Placebo Comparator

SUMMARY:
The ultimate objective of the proposed research is to improve the health-related quality of life of individuals with rheumatoid arthritis by reducing their risk of developing osteoporosis secondary to glucocorticoid therapy. The study has four specific aims.

Specific Aim 1: To obtain descriptive information concerning patients' knowledge, beliefs and behaviors with respect to osteoporosis and osteoporosis prevention.

Specific Aim 2: To identify factors that discriminate among patients in different stages of change with respect to each behavior of interest.

Specific Aim 3: To compare the effects of tailored versus generic educational materials on patient adherence to the ACR Guidelines for the Prevention of Glucocorticoid-Induced Osteoporosis.

Specific Aim 4: To determine if the effects of tailored educational materials are enhanced by concurrent feedback of information concerning patients' behavioral risk factor status to their physicians.

DETAILED DESCRIPTION:
Therapy with oral glucocorticoids often plays an important role in the management of rheumatoid arthritis (RA). The American College of Rheumatology (ACR) Ad Hoc Committee on Clinical Guidelines recently concluded that glucocorticoids are highly effective in relieving symptoms among people with active RA and that these medications may retard the rate of joint damage. Despite these obvious benefits, therapy with oral glucocorticoids is a well-established risk factor for osteoporosis, as highlighted by the recently published ACR Guidelines on the Prevention of Glucocorticoid-induced Osteoporosis. The ultimate objective of the proposed research is to improve the health-related quality of life of individuals with RA by reducing their risk of developing osteoporosis secondary to glucocorticoid therapy. The study has four specific aims: (1) to obtain descriptive information concerning patients' knowledge, beliefs and behaviors with respect to osteoporosis and osteoporosis prevention; (2) to identify factors that discriminate among patients in different stages of change with respect to each behavior of interest; (3) to compare the effects of tailored versus generic educational materials on patient adherence to the ACR Guidelines for the Prevention Glucocorticoid-induced Osteoporosis; and (4) to determine if the effects of tailored educational materials is enhanced by concurrent feedback of information concerning patients' behavioral risk factor status to their physicians. A sample of 273 patients with RA currently taking an oral glucocorticoid were recruited to participate in the study. Data were collected via mailed questionnaires and telephone interviews. The study used an experimental research design. Following baseline data collection, participants were randomly assigned to one of four experimental groups. Patients in one group received standard care only. Patients in the second group received generic educational materials about osteoporosis and osteoporosis prevention in addition to standard care. Patients in the third group received educational materials tailored to their stage in the behavior change process in addition to standard care. Finally, patients in the fourth group received the same tailored educational materials and care received by patients in the third group. In addition, each patient's physician received feedback concerning the patient's status with respect to behavioral risk factors for osteoporosis (e.g., inadequate calcium intake). Follow-up data were collected one year after baseline data collection. Variables assessed included: (1) behavior, (2) stage of change, (3) knowledge and counseling received concerning osteoporosis, (4) health beliefs, (5) physical health status, (6) osteoporosis risk factors, (7) background characteristics, and (8) information seeking. To accomplish the specific aims of the study, data will be analyzed using descriptive statistics, multivariate analysis of variance, and discriminant analyses.

ELIGIBILITY:
Inclusion Criteria:

* Meet American College of Rheumatology criteria for rheumatoid arthritis
* Taking an oral glucocorticoid equivalent to 5 mg/day of prednisone for at least one month prior to study entry
* Age 18 or older

Exclusion Criteria:

* Existing osteoporosis
* Pregnancy
* Breast feeding
* History of breast cancer
* Physician recommendation to limit calcium intake
* Class IV rheumatoid arthritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 273 (Actual)
Dates: Start 2001-07; Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Calcium Intake | One Year
Vitamin D Intake | One Year
Bone Mineral Density Testing | One Year
Use of prophylactic medications (e.g., bisphosphonates) | One Year

CONTACTS AND LOCATIONS:
Overall Officials: Susan J. Blalock, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill School of Pharmacy, Chapel Hill, North Carolina, United States

REFERENCES:
- [Result] Blalock SJ, Norton LL, Patel RA, Dooley MA. Patient knowledge, beliefs, and behavior concerning the prevention and treatment of glucocorticoid-induced osteoporosis. Arthritis Rheum. 2005 Oct 15;53(5):732-9. doi: 10.1002/art.21446. PMID 16208664